CLINICAL TRIAL: NCT00484484
Title: Efficacy of Low Analgesic Doses of Ketamine Associated With Opioids in Refractory Cancer Pain Treatment
Brief Title: Ketamine Associated With Opioids in Refractory Cancer Pain Treatment
Acronym: KETADOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Aurémie GUIMFACK, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P051048
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2007-06

CONDITIONS: Pain
Keywords: Cancer; Refractory pain; Uncontrolled pain; Ketamine; Uncontrolled cancer pain
MeSH Terms: conditions — Pain; Neoplasms; Pain, Intractable | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ketamine
  Interventions: Drug: Ketamine
- 2 (Experimental): Ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine

SUMMARY:
Long-term opioid therapy is commonly administered for the management of severe cancer pain. Increasing doses of opioids are titrated against effects until analgesia is achieved or intolerable adverse effects occur. Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has been reported to improve analgesia in patients with uncontrolled pain receiving high doses of opioids. This study aims at determining the effectiveness of ketamine as an adjuvant to opioids in relieving cancer pain.

DETAILED DESCRIPTION:
Main objective :

To show that low analgesic doses of ketamine associated with opioids better relieve refractory cancer pain than opioids without ketamine.

Secondary objectives :

* Determine whether ketamine use allows to reduce opioid consumption
* Evaluate the adverse effects of opioids-ketamine association versus opioids-placebo.

  100 patients are expected : 50 will be treated with opioids and ketamine ; 50 will be treated with opioids and a placebo.

Treatment will be administered for 4 days. Patients will be followed-up for 5 days.

Success is defined by a decrease of the daily pain score of 50 % after 4 days. The expected rate of success in the placebo group is 10 % whereas the expected rate of success in the ketamine group is 35 %.

Primary outcome (pain score on a 11-point numerical scale) will be evaluated everyday as well as secondary outcomes (patient and clinician global impression of change, opioid consumption, adverse reactions, patient satisfaction on pain relief, sleep interference score).

Vital parameters (cardiac frequency, respiratory frequency and arterial blood pressure) will be checked everyday, many times a day : every hour for the four hours after the beginning of the treatment and then, every four hours ; every hour for the two hours following a dose shift).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised cancer patients (informed and conscious of the cancer diagnostic)
* Undergoing opioid treatment for one month at least
* Refractory pain (score higher than 5 on an 11-point numerical pain rating scale)
* Ability to score pain on a numerical pain rating scale
* Patient written agreement

Exclusion Criteria:

* Ketamine contraindications
* Methadone or other NMDA-antagonist treatment
* Karnofsky index under 10
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Daily pain score on an 11-point numerical pain rating scale | after 4 days

SECONDARY OUTCOMES:
Patient Global Impression of Change Clinical Global Impression of Change Daily sleep interference score Patient satisfaction of pain relief Opioids consumption Adverse effects of ketamine-opioids association | during the 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie ROSTAING-RIGATTIERI, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint Antoine, Paris, France